CLINICAL TRIAL: NCT02781974
Title: The Effect of Exercise on Physical Function in Older Women With Osteoporosis and a History of Vertebral Fracture: A Randomized Controlled Trial
Brief Title: The Effect of Exercise on Physical Function in Older Women With Osteoporosis and a History of Vertebral Fracture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo Metropolitan University (Other)
Responsible Party: Principal Investigator, Brita Stanghelle, phd-student, Oslo Metropolitan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014/2050
Record Dates: First submitted 2016-05-18; First posted 2016-05-25 (Estimated); Last update posted 2019-03-08 (Actual); Status verified 2019-03

CONDITIONS: Osteoporosis; Vertebral Fractures
MeSH Terms: conditions — Osteoporosis; Spinal Fractures | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Intervention consists of strength and balance exercise in group sessions, twice a week for 12 weeks
  Interventions: Other: Exercise
- Control (No Intervention): Participants allocated in the control group are instructed to "live as usual"

INTERVENTIONS:
Other: Exercise — Strength and balance exercise in Groups, focusing on lower limb strength, back strength and static and dynamic balance
  Arms: Intervention

SUMMARY:
The study is a parallel-group single blinded randomized controlled trial, examining the effect of exercise on physical function in older women with osteoporosis and a history of vertebral fracture. The participants will randomly be assigned in a 1:1 ratio to the intervention group and the control group. The intervention will follow newly developed exercise recommendations for people with osteoporosis and vertebral fractures, which states the balance- and strength exercises should be performed at least twice a week. The intervention is a group exercise session circuit program lasting for 12 weeks. The participants will be tested at baseline, and followed up at 3 months and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Women over 65 years, living at home, able to walk with or without walking aids
* having osteoporosis verified by DXA scan (-2,5)
* at least one vertebral fracture, verified by X-ray

Exclusion Criteria:

* Health conditions that make it unsafe to exercise
* not able to understand and speak Norwegian adequately to participate in the intervention

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 149 (Actual)
Dates: Start 2016-01; Primary Completion 2018-10-12 (Actual); Study Completion 2018-10-12 (Actual)

PRIMARY OUTCOMES:
10 meter habitual walking speed | Up to 18 months

SECONDARY OUTCOMES:
Quality of life of participants assessed by the questionnaire Qualeffo 41 | Up to 18 months
Senior Fitness test | Up to 18 months
Functional reach | Up to 18 months
Four Square Step Test | Up to 18 months
Grip Strength | Up to 18 months
Short Form -36 | Up to 18 months
FES-1 | Up to 18 months
IPAQ-SF | Up to 18 months
Patient Specific Function Scale | Up to 18 months

CONTACTS AND LOCATIONS:
Locations (1):
- OsloMet - Oslo Metropolitan University, Oslo, Norway

REFERENCES:
- [Derived] Stanghelle B, Bentzen H, Giangregorio L, Pripp AH, Skelton DA, Bergland A. Physical fitness in older women with osteoporosis and vertebral fracture after a resistance and balance exercise programme: 3-month post-intervention follow-up of a randomised controlled trial. BMC Musculoskelet Disord. 2020 Jul 18;21(1):471. doi: 10.1186/s12891-020-03495-9. PMID 32682416
- [Derived] Stanghelle B, Bentzen H, Giangregorio L, Pripp AH, Skelton DA, Bergland A. Effects of a resistance and balance exercise programme on physical fitness, health-related quality of life and fear of falling in older women with osteoporosis and vertebral fracture: a randomized controlled trial. Osteoporos Int. 2020 Jun;31(6):1069-1078. doi: 10.1007/s00198-019-05256-4. Epub 2020 Jan 10. PMID 31925473
- [Derived] Stanghelle B, Bentzen H, Giangregorio L, Pripp AH, Bergland A. Associations between health-related quality of life, physical function and pain in older women with osteoporosis and vertebral fracture. BMC Geriatr. 2019 Nov 4;19(1):298. doi: 10.1186/s12877-019-1268-y. PMID 31684886
- [Derived] Stanghelle B, Bentzen H, Giangregorio L, Pripp AH, Bergland A. Effect of a resistance and balance exercise programme for women with osteoporosis and vertebral fracture: study protocol for a randomized controlled trial. BMC Musculoskelet Disord. 2018 Apr 3;19(1):100. doi: 10.1186/s12891-018-2021-y. PMID 29615028